CLINICAL TRIAL: NCT07326683
Title: Effect of Equivalent Dose of Oxycodone or Tegileridine on Patients Undergoing Gynecological Laparoscopic Hysterectomy
Brief Title: Clinical Study of Equivalent Doses of Oxycodone or Tegileridine on Patients Undergoing Gynecological Laparoscopic Hysterectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xin Chen (Other)
Collaborators: Second Affiliated Hospital of Hainan Medical College (Unknown)
Responsible Party: Sponsor-Investigator, Xin Chen, Associate Researcher,the Second Affiliated Hospital of Hainan Medical University, Hainan Medical College
Organization: Hainan Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUMU2H-TCOPOP-CN-2025; No.823RC592 (Other Grant/Funding Number: Hainan Provincial Natural Science Foundation of China)
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Total Laparoscopic Hysterectomy
Keywords: Tegileridine; Postoperative pain; Total Laparoscopic Hysterectomy; Oxycodone
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegileridine（T group） (Experimental): Around 20 minutes before the end of the operation, patients in the T group were given 0.01 mg/kg of Tegileridine(dissolved in 10 ml of 0.9% sodium chloride injection solution. This was administered via continuous infusion at a rate of 60 ml/h).
  Interventions: Drug: Tegileridine (tegileridine fumarate injection, IV)
- Oxycodone（O group） (Experimental): Around 20 minutes before the end of the operation, patients in the O group were given 0.06 mg/kg of Oxycodone(dissolved in 10 ml of 0.9% sodium chloride injection solution. This was administered via continuous infusion at a rate of 60 ml/h).
  Interventions: Drug: Oxycodone（Oxycodone Hydrochloride Injection，IV）

INTERVENTIONS:
Drug: Tegileridine (tegileridine fumarate injection, IV) — Tegileridine (tegileridine fumarate injection, IV) is a small-molecule μ-opioid receptor agonist with G-protein-biased signaling (relative to β-arrestin-2 recruitment), developed by Jiangsu Hengrui for postoperative analgesia. It is administered intravenously and was first approved in China in January 2024 for the treatment of moderate-to-severe pain after abdominal surgery; in this study, tegileridine is used as part of standardized multimodal analgesia according to protocol. In China it is regulated as a narcotic drug.
  Arms: Tegileridine（T group）
Drug: Oxycodone（Oxycodone Hydrochloride Injection，IV） — Oxycodone bitartrate is a dual opioid receptor agonist that is used in clinical settings. Oxycodone bitartrate injection is indicated for the relief of moderate to severe cancer pain. It can be administered alone or in combination with non-steroidal anti-inflammatory drugs to provide acute combined analgesia. In January 2021, Jiangsu Enhua Pharmaceutical submitted a marketing authorisation application for Oxycodone bitartrate injection to the National Medical Products Administration.The application has been accepted and approved.
  Arms: Oxycodone（O group）

SUMMARY:
This randomized, double-blind, controlled study aims to evaluate the efficacy and safety of Tegileridine or Oxycodone for postoperative analgesia in patients undergoing Total Laparoscopic Hysterectomy（TLH）. Subjects will be randomly assigned to receive an equivalent dose of intravenous Tegileridine or Oxycodone as part of a standard postoperative analgesia regimen. All patients will have access to rescue opioid analgesia according to the protocol. The primary objective is to determine if a single application of an equivalent dose of Tegileridine or Oxycodone can keep VAS scores at or below 3 during the anesthesia recovery phase. The secondary objectives are to compare cumulative opioid consumption within 48 hours postoperatively, time to first rescue analgesia, and the incidence rate of adverse events, such as nausea, vomiting, sedation, respiratory depression, pruritus, and constipation. Safety will be monitored throughout the study via predefined stop-and-report procedures. The study results will evaluate whether teglitazide provides a more effective, better-tolerated analgesic regimen for patients undergoing total laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing laparoscopic total abdominal hysterectomy with single-lumen endotracheal tube placement under general anaesthesia.
2. Females aged 18-65 years with a BMI of 18-28 kg/m²;
3. Normal mouth opening and head/neck mobility;
4. Preoperative American Society of Anesthesiologists (ASA) physical status classification of I-III and Mallampati airway classification of I or II;
5. Patients must also be scheduled for postoperative analgesia and have signed an informed consent form.

Exclusion Criteria:

1. Patients with allergies to the medications used in this study.
2. Patients with severe diseases of major organs, such as the heart, lungs or brain, including a history of acute myocardial infarction, cerebral infarction, asthma or chronic obstructive pulmonary disease;
3. Patients with severe liver or kidney dysfunction, or concomitant severe endocrine disorders such as poorly controlled hypertension, diabetes, hyperthyroidism or hypothyroidism.
4. Patients with a difficult airway, oropharyngeal/cervical anomalies, or a history of prior tracheostomy;
5. A history of prolonged sedative/analgesic use, substance abuse or opioid dependence;
6. Patients with neuropsychiatric disorders or impaired communication/comprehension abilities.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Success rate of postoperative pain management | After the surgery, before leaving the recovery room（Day 0）
  Following extubation during anaesthesia recovery after surgery, pain intensity was assessed at rest using a 10-cm visual analogue scale (VAS) by a blinded evaluator (with a minimum score of 0 indicating no pain and a maximum score of 10 indicating the most severe pain imaginable). Analgesia was recorded as successful when the VAS score was ≤3; otherwise, it was considered unsuccessful.

SECONDARY OUTCOMES:
Time of First Pressing of the PCIA | Within 48 hours after surgery
  Time of First Postoperative Pressing of the Patient-Controlled Intravenous Analgesia（PCIA） pump
Overall incidence of adverse reactions | Within 48 hours after surgery
  Incidence of Postoperative nausea and vomiting, hypotension, nasal congestion, dizziness, respiratory depression, delayed emergence from anesthesia, pruritus, muscle rigidity, convulsions, constipation, urinary retention, agitation during emergence, and convulsions.
Richmond Agitation and Sedation Scale(RASS) | Immediately before removal of the endotracheal tube (Postoperative Day 0).
  The research team assigns a RASS score (minimum -5 = unarousable, maximum +4 = combative; scores closer to 0 indicate an alert and calm state) by observing the patient immediately before tracheal extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology,the Second Affiliated Hospital of Hainan Medical University, Haikou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Apfel CC, Kranke P, Katz MH, Goepfert C, Papenfuss T, Rauch S, Heineck R, Greim CA, Roewer N. Volatile anaesthetics may be the main cause of early but not delayed postoperative vomiting: a randomized controlled trial of factorial design. Br J Anaesth. 2002 May;88(5):659-68. doi: 10.1093/bja/88.5.659. PMID 12067003
- [Result] Yu W, Wu X, Liu L, Long B, Tian Y, Ma C, Dong Y. The Median Effective Dose of One Intravenous Bolus of Oxycodone for Postoperative Analgesia After Myomectomy and Hysterectomy With Local Ropivacaine Wound Infiltration: An Up-Down Dose-Finding Study. Anesth Analg. 2020 Nov;131(5):1599-1606. doi: 10.1213/ANE.0000000000005011. PMID 33079884
- [Result] Wilder-Smith OH. Pre-emptive analgesia and surgical pain. Prog Brain Res. 2000;129:505-24. doi: 10.1016/S0079-6123(00)29037-7. No abstract available. PMID 11098714
- [Result] Kissin I. Preemptive analgesia. Anesthesiology. 2000 Oct;93(4):1138-43. doi: 10.1097/00000542-200010000-00040. No abstract available. PMID 11020772
- [Result] Kalso E. Oxycodone. J Pain Symptom Manage. 2005 May;29(5 Suppl):S47-56. doi: 10.1016/j.jpainsymman.2005.01.010. PMID 15907646